CLINICAL TRIAL: NCT04926324
Title: A Phase 1b/2 Trial of Preoperative Niraparib, Dostarlimab, and Hypofractionated Radiotherapy for the Treatment of Locally-advanced Rectal Cancers.
Brief Title: A Safety Study Adding Niraparib and Dostarlimab to Radiation Therapy for Rectal Cancers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor terminated
Sponsor: University of Iowa (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Kellie Bodeker, Associate Director of Theranostics Research, University of Iowa
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202103459
Record Dates: First submitted 2021-06-08; First posted 2021-06-15 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Rectal Neoplasms; Rectal Neoplasm Malignant
Keywords: niraparib; dostarlimab; radiation therapy; total neoadjuvant therapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — niraparib; dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (starting) (Experimental): niraparib, 100 mg orally once daily for up to 12 weeks dostarlimab, 500 mg infused (IV) once every 3 weeks for up to 12 weeks radiation therapy, 5 Gray (Gy) per day for 5 consecutive days
  Interventions: Drug: Niraparib; Drug: Dostarlimab; Radiation: Short course radiation
- Cohort 2 (Experimental): niraparib, 200 mg orally once daily for up to 12 weeks dostarlimab, 500 mg infused (IV) once every 3 weeks for up to 12 weeks radiation therapy, 5 Gray (Gy) per day for 5 consecutive days
  Interventions: Drug: Niraparib; Drug: Dostarlimab; Radiation: Short course radiation

INTERVENTIONS:
Drug: Niraparib — Niraparib is a drug FDA-approved for use in maintenance treatment of adults with advanced ovarian cancer, fallopian tube cancer, or primary peritoneal cancer.
  Other Names: Zejula
Drug: Dostarlimab — Dostarlimab, sold under the brand name Jemperli, is a monoclonal antibody medication used for the treatment of endometrial cancer.
  Other Names: Jemperli
Radiation: Short course radiation — Participants will be treated with intensity modulated radiation therapy (IMRT) or volumetric modulated arc therapy (VMAT) to minimize mean dose to femoral, pelvic, and lumbar bone marrow. The entire mesorectum will be treated to a total dose of 25 Gy.
  Other Names: IMRT; VMAT

SUMMARY:
This clinical trial is designed to determine the maximum tolerated dose of niraparib when combined with dostarlimab and hypofractionated radiation for locally advanced rectal cancer. Once this is determined, this dose will be tested to identify what impact it has on the tumor as well as patient reported outcome measures.

DETAILED DESCRIPTION:
Standard of care therapy for resectable locally advanced rectal cancer includes pelvic radiation (short or long course), chemotherapy, and (if indicated) surgery.

In this study, participants will:

* Take niraparib by mouth once daily for up to 12 weeks.
* Receive radiation therapy once daily for five days (Monday through Friday).
* Receive intravenous (IV) dostarlimab once every three weeks for up to 12 weeks.
* Provide feedback about how they feel and their quality of life. This is done through short surveys as well as discussing with the study team.
* Undergo a sigmoidoscopy (i.e. scope of the tumor) and biopsy about halfway through treatment
* Provide tumor tissue and blood samples for analysis

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to provide independent informed consent; legally authorized representative consent and/or power-of-attorney is not allowed.
* Age at least 18 years at the time of study drug administration
* Resectable locally advanced rectal cancer (i.e., T3 to T4 or T1-T4 with N1-2 M0).
* Recommended to receive total neoadjuvant therapy consisting of preoperative radiation therapy followed by systemic FOLFOX chemotherapy
* Adequate performance status (ECOG of 0 or 1; or KPS of >70).
* Agree to adhere to lifestyle considerations throughout study duration
* Agree to not donate blood during the study or for 90 days after the last dose of study treatment.

Exclusion Criteria:

* Absolute neutrophil count < 1,500 cells /µL
* Platelets < 100,000 cells/µL
* Hemoglobin <9 g/dL
* Serum creatinine > 1.5 x upper limit of normal (ULN) or calculated creatinine clearance 60mL/min using the Cockcroft-Gault equation
* Total bilirubin > 1.5 x ULN (>2.0 x ULN in patients with known Gilberts syndrome) or direct bilirubin > 1 x ULN
* Aspartate aminotransferase and alanine aminotransferase > 2.5 x ULN
* International normalized ratio (INR) or prothrombin time (PT) >1.5× ULN unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin (PTT) is within therapeutic range of intended use of anticoagulants.
* Activated partial thromboplastin time (aPTT) >1.5× ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Uncontrolled arterial hypertension, i.e. systolic BP > 140 mmHg, diastolic BP > 90 mmHg.
* Platelet transfusion ≤ 4 weeks prior to initiating protocol therapy.
* Presence of any M1 metastatic lesions.
* Prior pelvic radiotherapy
* Indication for total neoadjuvant therapy or alternative radiation regimen
* Recommended to receive a chemotherapy regimen other than FOLFOX chemotherapy. CapeOX (oral xeloda plus oxaliplatin) is an acceptable alternative as it contains the core fluoropyrimidine + oxaliplatin backbone.
* Indication for alternative radiation dose or fractionation regimen.
* Active Crohn's disease or another inflammatory bowel disease
* Any T or N stage disease that is deemed unresectable by colorectal surgery without neoadjuvant therapy
* Prior anti-PD-L1 therapy, PARPi therapy, or known germline BRCA-1/2 mutation as patients with germline BRCA-1/2 mutations have an increased risk of severe normal tissue injury to combination radiation and PARP inhibition.
* Received a live vaccine within 14 days of initiating protocol therapy.
* Received colony stimulating factors (e.g., granulocyte colony-stimulating factor, granulocyte macrophage colony stimulating factor, or recombinant erythropoietin) within 4 weeks prior to Day 1 of protocol therapy.
* Major surgery within 3 weeks prior to Day 1 of protocol therapy (participant must recover from any surgical effects).
* Investigational therapy ≤ 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, prior to Day 1 of protocol therapy.
* Known hypersensitivity to niraparib and dostarlimab components or excipients.
* Known grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment.
* Known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
* Diagnosis, detection, or treatment of another type of cancer ≤ 2 years prior to initiating protocol therapy (except basal or squamous cell carcinoma of the skin and cervical cancer that has been definitively treated).
* Known history of ≥ grade 3 immune-related AE with prior immunotherapy, with the exception of non-clinically significant lab abnormalities.
* Diagnosis of immunodeficiency or has received systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to initiating protocol therapy.
* Patients with known HIV who have documented detectable viral load or patients with a documented undetectable viral load and a CD 4 count < 350 cells within 6 months of study treatment day
* Known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [qualitative] is detected).
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* History of interstitial lung disease.
* Active or uncontrolled infection necessitating hospitalization or treatment delay.
* Known serious, uncontrolled medical disorder or nonmalignant systemic disease that preclude eligibility to undergo low anterior resection (LAR). Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, or any psychiatric disorder that prohibits obtaining informed consent
* Pregnancy. Participant must have a negative serum pregnancy test within 72 hours prior to taking study treatment if of childbearing potential and agrees use a highly effective method of contraception from screening through 180 days after the last dose of niraparib and after the last dose of dostarlimab, or is of nonchildbearing potential. Nonchildbearing potential is defined as follows (by other than medical reasons):

  1. ≥ 60 years of age
  2. Post-hysterectomy. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound.
* Actively breastfeeding. Participant must agree to not breastfeed during the study or for 8 weeks after the last dose of study treatment.
* Declines to use a highly effective method of contraception (see Section 5.2.1 for a list of acceptable birth control methods). Eligible patients must agree to highly effective methods of contraception starting with the first dose of study treatment through 180 days after the last dose of niraparib and dostarlimab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-12-26 (Actual)

PRIMARY OUTCOMES:
Determination of recommended phase 2 niraparib dose | From treatment day 1 for up to 16 weeks.
  The recommended dose will be determined by incidence of dose limiting toxicities.
Determination of the clinical complete response rate | 8
  Clinical evaluation of the tumor by both flexible sigmoidoscopy and pelvic MRI

SECONDARY OUTCOMES:
Determine overall survival (OS) | Time (measured in days) until death from any cause, up to 20 years post-treatment.
  Time from treatment day 1 to death from any cause
Determine progression free survival (PFS) | From treatment day 1 to disease progression, up to 15 years post-treatment
  Time (measured in days) to documented disease progression in imaging as described by the RECIST criteria.
Determine metastasis free survival | From treatment day 1 to disease progression or death, up to 20 years post-treatment.
  Time (measured in days) to documented disease progression outside of the pelvis or death from any cause.
Determine local recurrence free survival | From treatment day 1 to disease progression or death, up to 20 years post-treatment.
  Time (measured in days) to disease progression within the pelvis or death from any cause.
Determine ostomy free survival | From treatment day 1 up to 20 years post-treatment.
  Time (measured in days) to receipt of permanent ostomy or death from any cause.
Determine objective response rate | 3 months post-radiation
  Objective response rate, measured using the standardized RECIST criteria, is a reflection of complete tumor response and partial tumor response. The
Determination of the pathologic complete response | At surgery; up to 1 year post-treatment
  Absence of viable tumor in the primary tumor bed and all regional nodes in patients recommended to undergo surgical resection regardless of response to neoadjuvant therapy.
Determination of the organ preservation rate | From treatment day 1 up to 15 years post-treatment
  Organ perservation defined as day 1 therapy to receipt of rectal resection for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Kellie Bodeker, Ph.D., Principal Investigator — University of Iowa
Locations (1):
- Holden Comprehensive Cancer Center at the University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be released publicly as per participant consent and IRB approval. Individual researchers should contact the research team for data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study protocol and informed consent will be shared after primary completion. Statistical analysis plan will be shared with results reporting.
Access Criteria: An IRB-stamped signed usage agreement will be required in addition to a data sharing agreement between the academic centers.

REFERENCES:
- [Background] Seyedin SN, Hasibuzzaman MM, Pham V, Petronek MS, Callaghan C, Kalen AL, Mapuskar KA, Mott SL, Spitz DR, Allen BG, Caster JM. Combination Therapy with Radiation and PARP Inhibition Enhances Responsiveness to Anti-PD-1 Therapy in Colorectal Tumor Models. Int J Radiat Oncol Biol Phys. 2020 Sep 1;108(1):81-92. doi: 10.1016/j.ijrobp.2020.01.030. Epub 2020 Feb 6. PMID 32036006

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT04926324/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT04926324/ICF_001.pdf